CLINICAL TRIAL: NCT01037166
Title: A Phase II Study in Japan of the Safety And Antiviral Activity of Entecavir (BMS-200475) in Adults With Chronic Hepatitis B With Incomplete Response to Current Lamivudine Therapy
Brief Title: Study in Japan of the Safety And Antiviral Activity in Adults With Chronic Hepatitis B Current Lamivudine Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI463-052
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Entecavir (0.5 mg) (Experimental)
  Interventions: Drug: Entecavir
- Entecavir (1mg) (Experimental)
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — Tablet, P.O., 0.5 mg or 1mg, once daily, 52 weeks
  Other Names: Baraclude; BMS-200475

SUMMARY:
The objectives are to demonstrate that entecavir has antiviral activity undetectable HBV DNA measured, the Roche AmplicorTM PCR at Week 48, and to assess the safety and the pharmacokinetic of entecavir in Japanese patients with hepatitis B who have an incomplete response to current lamivudine therapy

ELIGIBILITY:
Inclusion Criteria:

* Documentation of chronic hepatitis B infection by ALL of the following:

  1. Positive for HBsAg OR, negative for IgM core antibody and confirmation of chronic hepatitis B on liver biopsy
  2. Patient who have received lamivudine therapy for 24 weeks or more, or patient who have documented YMDD mutation or other lamivudine-resistant mutation while on lamivudine
  3. Documented HBV Viremia ≥ 10*5: copies/mL
* ALT in the range of 1.3 to 10 x ULN
* Subjects must have well-compensated liver disease a) value

Exclusion Criteria:

-

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2002-12; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
To assess the safety (the incidence of clinical adverse events and discontinuations due to adverse events) | Week 52 (end of dosing) plus 5 days
To assess the proportion of subjects with reduction in HBV DNA by ≥ 2 log10 or to undetectable level (< 400 copies/mL) | at Week 48

SECONDARY OUTCOMES:
Mean change from baseline in the log*10* HBV DNA measured by PCR assay for each entecavir dose (0.5 and 1 mg) at Week 48 | Baseline, Week 48
Proportion of subjects who achieve undetectable HBV DNA (<400 copies/mL) by PCR assay at Week 48 | Week 48
Proportion of subjects HBeAg-positive at baseline who have loss of HBeAg from serum at Week 48 | Week 48
Proportion of subjects HBeAg-positive at baseline who achieve seroconversion (loss of HBeAg and appearance of HBeAb) at Week 48 | Week 48
Proportion of subjects with abnormal ALT at baseline who achieve normalization of serum ALT (<1.25 x ULN) at Week 48 | Week 48
Proportion of subjects HBeAg-positive at baseline who have complete response (undetectable HBV DNA levels by PCR assay, negative for HBeAg and normal serum ALT) at Week 48 | Week 48
Proportion of subjects HBeAg-negative at baseline who have undetectable HBV DNA levels by PCR assay, remain negative for HBeAg and normal serum ALT at Week 48 | Week 48
Proportion of subjects w/ histological improvement in liver (improvement in necroinflammatory score (≥2 points decrease, Knodell HAI3 score) & no worsening of fibrosis (≥1 point increase, Knodell fibrosis score) at Wk 48 liver biopsy compared to baseline | Baseline, Week 48
Changes in liver histology as assessed by the New Inuyama Classification for histological assessment of chronic hepatitis | Week 52
Relationship between HBV isolates (genotypes A,B,C, etc.) at baseline and antiviral activity | Week 48, or at end of dosing (up to Week 52)
Incidence of resistance mutations of HBV isolates in subjects who have a rise in HBV DNA (by ≥1 log above the nadir for that subject) while on study drug. | Week 48, or at end of dosing (up to Week 52)
Mutation of HBV DNA polymerase at Week 48 from baseline | Baseline, Week 48
Plasma concentrations of entecavir at selected time points during the treatment period | pre-dosing, Week 2 or 4, Week 12, Week 24 and Week 36
Population pharmacokinetic assessment of entecavir developed from concentration-time data obtained from healthy subjects | pre-dosing, Week 2 or 4, Week 12, Week 24 and Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- Japan (15):
  - Local Institution, Aichi-Gun, Aichi-ken
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Chiba, Chiba
  - Local Institution, Kurume, Fukuoka
  - Local Institution, Ogaki-Shi, Gifu
  - Local Institution, Asahikawa-Shi, Hokkaido
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Akashi-Shi, Hyōgo
  - Local Institution, Morioka, Iwate
  - Local Institution, Kyoto, Kyoto
  - Local Institution, Sendai, Miyagi
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Minato-Ku, Tokyo
  - Local Institution, Musashino-Shi, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo

REFERENCES:
- [Background] Suzuki F, Toyoda J, Katano Y, Sata M, Moriyama M, Imazeki F, Kage M, Seriu T, Omata M, Kumada H. Efficacy and safety of entecavir in lamivudine-refractory patients with chronic hepatitis B: randomized controlled trial in Japanese patients. J Gastroenterol Hepatol. 2008 Sep;23(9):1320-6. doi: 10.1111/j.1440-1746.2008.05455.x. Epub 2008 Jun 28. PMID 18554238
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx